CLINICAL TRIAL: NCT06375473
Title: Treatment of Irinotecan Hydrochloride Liposome Injection II in China: a Real World Study of Pancreatic Cancer Patients
Acronym: MA-PC-RWS-011
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MA-PC-RWS-011
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
Keywords: real word study, irinotecan hydrochloride liposome injection II, pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Perioperative cohort: Irinotecan liposome II combination therapy regimen for perioperative patients
  Interventions: Drug: Irinotecan liposome II combination therapy regimen
- First line cohort: Irinotecan liposome II combination therapy regimen for first line advanced patients
- Second line cohort: Irinotecan liposome II combination therapy regimen for second line advanced patients
- Late stage third line and above cohort: Irinotecan liposome II combination therapy regimen for third line and above advanced patients

INTERVENTIONS:
Drug: Irinotecan liposome II combination therapy regimen — Irinotecan liposome II combination therapy regimen
  Groups: Perioperative cohort

SUMMARY:
This study is a multi-center observational study.The start time for data collection is May 1, 2024. Patients' baseline and treatment data will be collected under informed concent. The purpose of this case registry study was to evaluate the safety and efficacy of irinotecan hydrochloride liposome injection II based therapy in Chinese patients with pancreatic cancer in the real world by collecting, understanding, and analyzing the etiology, clinical features, treatment pattern, treatment outcomes, and pharmacoeconomics changes in pancreatic cancer patients receiving this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic ductal adenocarcinoma diagnosed by pathology or imaging;
* Age ≥18 years old, male or female;
* Patients receiving treatment based on irinotecan hydrochloride liposome injection II;
* The subjects voluntarily joined the study and signed the informed consent.

Exclusion Criteria:

* Confirmed pregnant or lactating women;
* The researchers determined that other conditions were not suitable for inclusion in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients in China
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
rwTEAE | 3 years
  real word treatment emergent adverse event

SECONDARY OUTCOMES:
OS | 3 years
  real word overall survival
PFS | 3 years
  real word progression free survival
ORR | 3 years
  real word objective response rate
TTP | 3 years
  real word time to progression
DCR | 3 years
  real word disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Taiping Zhang, doctor, Principal Investigator — Peking Union Medical College Hospital, Beijing, China; Liwei Wang, doctor, Principal Investigator — Renji Hospital, Shanghai, China
Locations (10):
- China (10):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Peking Unicersity First Hospital, Beijing
  - Henan Provincial People's Hospital, Henan
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji，Hospital, Shanghai
  - Wuhan Union Hospital of China, Wuhan